CLINICAL TRIAL: NCT05432726
Title: Prediction of Chemotherapy Toxicity and Survival in Elderly Cancer Patients by Using CARG Score (Cancer and Aging Research Group Score)
Brief Title: Prediction of Chemotherapy Toxicity and Survival in Elderly Cancer Patients by CARG Score
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Donia Hussein Abd Elhamed, Assistant Lecturer, Assiut University
Other Study IDs: CARG Score in Elderly Patients
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Solid Tumors ,Adults
Keywords: CARG score - Elderly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elderly patients: Elderly patients (aged ≥65 year's old) planned to receive first-line chemotherapy for advanced solid tumor malignancies, presenting to the clinical oncology department, Assiut University Hospitals, Assiut, Egypt.
  Interventions: Other: calculating CARG score

INTERVENTIONS:
Other: calculating CARG score — Before the initiation of chemotherapy, study participants will complete the GA questions included in the CARG toxicity score.
  Total risk score will be calculated ranging from 0 (lowest toxicity risk) to 19 (highest toxicity risk), incorporates measures of functional status such as fall history, hearing problems, physical capabilities, performance status as well as objective measures including age, gender, height, weight, cancer type, type and dose of chemotherapy, hemoglobin, and creatinine clearance.
  CARG score will be stratified as low (score 0-5), intermediate (score 6-9) and high risk (score 10-19).
  Chemotherapy-related toxicities will be assessed and graded as per the NCI-CTCAE, version 5.0.
  Hospitalizations due to AEs during first-line chemotherapy will be collected.
  Subsequent changes in chemotherapy dosage, treatment delays, and treatment discontinuation due to adverse effects as well as mortality rate after treatment will also be monitored.

SUMMARY:
Prediction of chemotherapy toxicity and survival in elderly (aged ≥65 years old) patients with advanced solid tumors receiving systemic chemotherapy by using CARG risk score.

DETAILED DESCRIPTION:
Elderly patients (age ≥65 years) with cancer represent a growing proportion of patients in oncology clinical practice, primarily due to increasing life-spans as well as medical progress contributing to decreased morbidity and mortality from other causes.

Treatment decision-making for elderly patients with advanced cancer is often more complex than decision-making in younger cancer patients. The elderly population is heterogeneous in terms of their overall health status beyond their cancer diagnosis.

The risk of severe chemotherapy toxicity is one of the most important factors oncologists consider when recommending a treatment plan, and in elderly patients with advanced cancers, 25% to 60% of patients are treated with a planned dose reduction for their first chemotherapy cycle. These dose reductions are usually made on the basis of chronologic age and ECOG performance status, variables well known to be poor predictors of chemotherapy toxicity risk and tolerability of treatment.

Clinical prediction tools provide physicians with more accurate means for identifying patients who are at low or high risk of adverse outcomes.

The cancer Aging Research Group (CARG) risk score, developed by Hurria and colleagues, is a validated geriatric assessment tool that predicts for significant chemotherapy-related toxicities (grades 3-5) in older North American adults aged ≥65 years starting on chemotherapy.

The CARG score uses 5 key geriatric assessment (GA) domains, selected laboratory test values, age, tumor type, and treatment intensity to categorize patients into 3 risk groups for severe chemotherapy toxicity (grade 3-5): low risk (score 0-5; 30% grade 3-5 toxicity), medium risk (score 6-9; 52%), or high risk (score ≥10; 83%).

The CARG risk score has been validated in other countries and in specific tumour sites to varying degrees. It is included in ASCO Guideline and NCCN guidelines for Geriatric Oncology to predict severe chemotherapy-related toxicity. However its applicability in Egyptian patients is unknown as geriatric assessment is not routinely used for elderly patients.

The investigators may provide an evidence for validating the CARG risk score in Elderly patients with advanced solid tumors receiving systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥65 years.
* Sex: male, female.
* ECOG performance status 0,1,2
* Type of malignancy: solid tumor malignancies planned for systemic chemotherapy alone.
* Stage: Advanced stage (metastatic first line, recurrent, unresectable locally advanced).
* Type of Systemic therapy: chemotherapy alone not combined with immunotherapy or radiotherapy.
* Able to comprehend and complete questionnaire.

Exclusion Criteria:

* Receiving concurrent radiotherapy or immunotherapy.
* ECOG performance status >2.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (aged ≥65 year's old) planned to receive first-line chemotherapy for advanced solid tumor malignancies, presenting to the clinical oncology department, Assiut University Hospitals, Assiut, Egypt, from june 2022 to june 2023.
Sampling Method: Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2022-07-20 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Prediction of grade 3-5 chemotherapy toxicity risk in elderly patients (aged ≥65 years old) with advanced solid tumors by measurement of CARG risk score (Cancer and Aging Research Group). | 6 months follow up in first line chemotherapy in the advanced setting

SECONDARY OUTCOMES:
Correlation of the physician measured ECOG PS with grade 3-5 toxicities. | 6 months follow up in first line chemotherapy in the advanced setting
Correlation between the CARG score and 2 year PFS (progression free survival). | 2 years
  it will be measured from the time from start of first-line chemotherapy to disease progression or, censored at last clinic visit)
Correlation between the CARG score and 2 year OS (overall survival). | 2 years
  it will be measured from the start of chemotherapy to death or censored at the last clinic visit

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Moth EB, Kiely BE, Stefanic N, Naganathan V, Martin A, Grimison P, Stockler MR, Beale P, Blinman P. Oncologists' perceptions on the usefulness of geriatric assessment measures and the CARG toxicity score when prescribing chemotherapy for older patients with cancer. J Geriatr Oncol. 2019 Mar;10(2):210-215. doi: 10.1016/j.jgo.2018.11.004. Epub 2018 Nov 28. PMID 30503312
- [Result] Ortland I, Mendel Ott M, Kowar M, Sippel C, Jaehde U, Jacobs AH, Ko YD. Comparing the performance of the CARG and the CRASH score for predicting toxicity in older patients with cancer. J Geriatr Oncol. 2020 Jul;11(6):997-1005. doi: 10.1016/j.jgo.2019.12.016. Epub 2020 Jan 9. PMID 31928942
- [Result] Nishijima TF, Deal AM, Williams GR, Sanoff HK, Nyrop KA, Muss HB. Impact of the Cancer and Aging Research Group score and treatment intensity on survival and toxicity outcomes in older adults with advanced noncolorectal gastrointestinal cancers. Cancer. 2022 May 15;128(10):1929-1936. doi: 10.1002/cncr.34135. Epub 2022 Feb 11. PMID 35147991
- [Result] DuMontier C, Sedrak MS, Soo WK, Kenis C, Williams GR, Haase K, Harneshaug M, Mian H, Loh KP, Rostoft S, Dale W, Cohen HJ. Arti Hurria and the progress in integrating the geriatric assessment into oncology: Young International Society of Geriatric Oncology review paper. J Geriatr Oncol. 2020 Mar;11(2):203-211. doi: 10.1016/j.jgo.2019.08.005. Epub 2019 Aug 23. PMID 31451439
- See also: Cancer Aging Research Group (CARG) score in older adults undergoing curative intent chemotherapy: a prospective cohort study — https://bmjopen.bmj.com/content/11/6/e047376.abstract